CLINICAL TRIAL: NCT01259141
Title: The Optimization of Mycoplasm Pneumonia Antibiotic Therapy: Multi-centre, Prospective, Randomized Controlled Study
Brief Title: The Optimization of Mycoplasm Pneumonia Antibiotic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Bin Cao, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MP201011
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Mycoplasma Pneumonia
Keywords: macrolide- resistant Mycoplasma pneumoniae,; Mycoplasm pneumonia antibiotic therapy
MeSH Terms: conditions — Pneumonia, Mycoplasma | interventions — Moxifloxacin; Cephalosporins; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moxifloxacin (Experimental)
  Interventions: Drug: Moxifloxacin
- Cephalosporins and azithromycin (Experimental)
  Interventions: Drug: Cephalosporins and azithromycin

INTERVENTIONS:
Drug: Moxifloxacin — 0.4 Qd for 7days
  Arms: Moxifloxacin
Drug: Cephalosporins and azithromycin — cefuroxime 1.5 bid for 7 days plus azithromycin 0.5 qd for 7 days
  Arms: Cephalosporins and azithromycin

SUMMARY:
Mycoplasma pneumoniae, an important pathogen of community acquired pneumonia,are becoming more and more resistant to macrolide. The study aim is to optimize anti-infection therapy.

DETAILED DESCRIPTION:
Mycoplasma pneumoniae was one of important atypical pathogens of community acquired pneumonia. As lack of cell wall, β-lactam medicines were invalid, however, macrolides, tetracyclines and quinolones were effective. But from 2001, many countries reported macrolide- resistant Mycoplasma pneumoniae. Typically, erythromycin was first-line antibiotic medicine. With the resistance increasing, Mycoplasm pneumonia treatment will become more and more difficult. Thus, optimization of Mycoplasm pneumonia antibiotic therapy is very important.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed community acquired pneumonia
2. 60ys≥age≥18 ys
3. Respiratory symptom (cough accompanied by little or no sputum)
4. New infiltration showed by chest radiology(x-ray or CT)
5. Lung signs was not obvious
6. White blood cell<10,000/mm3
7. Without underlying diseases or mild

Exclusion Criteria:

1. Age<18ys or >60ys
2. Pregnancy or breast-feeding
3. Over one week after the onset of symptoms
4. HIV infection
5. Recent 90-day hospitalized history(length of stay greater than 2 days)
6. Live in nursing homes or rehabilitation hospitals
7. Taken macrolides or quinolones medicines before enrollment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 208 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Time to resolution of fever (defined as the period from start of study-drug to relief of fever) | one month
  usually duration of fever is about one to two weeks
Time to resolution of fever (defined as the period from onset to relief of fever) | one month
  usually duration of fever is about one to two weeks

SECONDARY OUTCOMES:
Time to resolution of respiratory symptoms(defined as the period from start of study-drug to relief of symptoms) | one year
Time to resolution of respiratory symptoms(defined as the period from onset to relief of symptoms) | one year
Proportion of antibiotics change | one year
Duration of antibiotics | one year
Proportion of resolution of fever after antibiotics therapy for 24 hours | one year
Proportion of resolution of fever after antibiotics therapy for 72 hours | one year
Antibiotic-related adverse reaction | one year

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cao, Doctor, Study Chair — Capital Medical University affiliated Beijing Chaoyang Hospital, Beijing Respiratory Medicine Insititute
Locations (1):
- Capital Medical University affiliated Beijing Chaoyang Hospital, Beijing Respiratory Medicine Insititute, Beijing, Beijing Municipality, China